CLINICAL TRIAL: NCT04815304
Title: Clinical Features of Severe Acute Respiratory Syndrome Coronavirus 2 Patients Admitted to the Intensive Care Units of Academic Hospital of L'Aquila (Italy)
Brief Title: Clinical Features of COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Medical Doctor, San Salvatore Hospital of L'Aquila
Other Study IDs: 26100/21
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Covid19; Acute Respiratory Distress Syndrome; Ventilatory Failure
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Hypoventilation | interventions — Blood Gas Analysis; Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: peripheral lymphocytes subsets — The data were collected during the first and the second wave of epidemic in COVID-19 patients with acute respiratory distress syndrome. At the moment of hospitalization, at the moment of intensive care unit admission and during the in intensive care unit staying, the following data were collected: peripheral lymphocyte subsets were measured by multiple-color flow cytometry, chest computed tomography and ultrasonography scans (lung ultrasound score, diaphragmatic thickness and motion), arterial blood gas analysis parameters (pH, partial pressure of carbon dioxide, partial pressure of oxygen, concentration of hydrogen carbonate, base excess, and arterial oxygen saturation ), and pain assessed by using numeric rating scale. Macroscopic and microscopic hypopharynx and larynx damages were also evaluated by video-laryngoscopy and light miscoscopy.
  Other Names: Chest computed tomography; Chest ultrasonography scan; arterial blood gas analysis; pain

SUMMARY:
The data were retrospectively collected during the first and the second wave of epidemic in COVID-19 patients with Severe Acute Respiratory Syndrome Coronavirus 2, at the moment of intensive care unit admission and during the in intensive care unit staying.

DETAILED DESCRIPTION:
At the moment of intensive care unit admission and during the in intensive care unit staying, the following data were collected: peripheral lymphocyte subsets were measured by multiple-color flow cytometry, chest computed tomography and ultrasonography scans, arterial blood gas parameters (pH, partial pressure of carbon dioxide, partial pressure of oxygen, concentration of hydrogen carbonate, base excess, and arterial oxygen saturation), and pain assessed by using numeric rating scale.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients
* Acute respiratory distress syndrome
* needing of ventilatory support

Exclusion Criteria:

* asymptomatic COVID-19 patients
* few symptoms
* mild symptoms
* without needing of ventilatory support

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data were collected during the first and the second wave of epidemic in COVID-19 patients with acute respiratory distress syndrome
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Peripheral lymphocyte subsets | Change from date of hospitalization until the date of hospital discharge or date of death from any cause, whichever came first, assessed at 60 weeks
  Peripheral lymphocyte subsets were measured by multiple-color flow cytometry,

SECONDARY OUTCOMES:
Chest computed tomography | From date of hospitalization until the date of hospital discharge or date of death from any cause, whichever came first, assessed every 10 days up to 60 weeks
  A chest computed tomography performed to assess lung damage
Chest ultrasonography | From date of hospitalization until the date of hospital discharge or date of death from any cause, whichever came first, assessed every day up to 60 weeks
  Lung ultrasound score (sum of points in all 12 regions and ranges from 0 to 36; 0 points-presence of lung sliding with A lines or one or two isolated B lines; 1 point-moderate loss of lung aeration with three or four B lines (septal rockets); 2 points-severe loss of lung aeration with five or more B lines (glass rockets); and 3 points-presence of a hypoechoic poorly defined tissue characterized by consolidation)
Pain assessment | From date of hospitalization until the date of hospital discharge or date of death from any cause, whichever came first, assessed every day up to 60 weeks
  Pain assessed by using numeric rating scale (the 11-point numeric scale ranges from '0' representing one pain extreme [e.g. "no pain"] to '10' representing the other pain extreme [e.g. "pain as bad as you can imagine" or "worst pain imaginable])
Upper airway damages | From date of hospitalization until the date of hospital discharge or date of death from any cause, whichever came first, assessed every day up to 60 weeks
  Macroscopic and microscopic hypopharynx and larynx damages evaluated by video-laryngoscopy and light microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Franco Marinangeli, MD, Study Chair — ASL 1 Avezzano Sulmona L'Aquila
Locations (1):
- San Salvatore Academic Hospital, L’Aquila, Italy